CLINICAL TRIAL: NCT05570019
Title: Evaluation of Tissue Perfusion in Patients With Lower Extremity Peripheral Arterial Disease
Brief Title: Evaluation of Tissue Perfusion in Peripheral Arterial Disease (EVTI-PAD)
Acronym: EVTI-PAD
Status: Recruiting | Type: Observational
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Other Study IDs: 1440/2021
Record Dates: First submitted 2022-08-29; First posted 2022-10-06 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Peripheral Arterial Disease; Chronic Limb-Threatening Ischemia; Critical Limb Ischemia
Keywords: Tissue perfusion; Peripheral arterial disease; Critical limb threatening ischemia; Critical limb ischemia; Fluorescence angiography; Fluorescence imaging; Indocyanine green; Microcirculation
MeSH Terms: conditions — Peripheral Arterial Disease; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Revascularization — Open surgery (arterial endarterectomy with or without bypass surgery) and/or angioplasty (with or without stent placement)

SUMMARY:
In this prospective single-center observational study, arterial perfusion in patients with lower limb peripheral arterial disease will be assessed with standard diagnostic tools (toe pressure, trans-cutaneous oxygen pressure, ankle-brachial index and fluorescence angiography) before and after standard revascularization procedures (open surgery and/or angioplasty).

DETAILED DESCRIPTION:
Arterial perfusion is an important parameter for the capacity of wound healing in patients with peripheral arterial disease (PAD). Quantifying tissue perfusion in affected patients can help in deciding whether further revascularization is necessary to achieve wound healing and limb salvage. Not only in PAD patients with ulceration, but also in patients with rest pain or life-style limiting claudication, the measurement of arterial perfusion before and after revascularization could influence further treatment regarding surgical/interventional procedures as well as medical treatment. Digital subtraction angiography (DSA) is the gold standard for the evaluation of peripheral arterial outflow and for quality assessment after revascularization. However, angiography only displays the larger arteries and not tissue perfusion itself, which is crucial for wound healing. In this study, the change of tissue perfusion measured with the different standard diagnostic tools (toe pressure, trans-cutaneous oxygen pressure, ankle-brachial index and fluorescence angiography) before and after standard revascularization procedures will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

- patients with symptomatic peripheral arterial disease (Rutherford categories 3-6) requiring revascularization.

Exclusion Criteria:

* patients younger than 18 years
* patients unable to give consent without legal guardians
* iodine allergy
* hyperthyroidism
* allergy to indocyanine green
* Glomerular filtration rate <30ml/min/1.73m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic peripheral arterial disease (Rutherford categories 3-6) requiring revascularization procedures (open surgery and/or angioplasty).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Transcutaneous oxygen pressure | Pre-procedural, post-procedural (within 5 days) and 3 months after the index procedure
  Change in transcutaneous oxygen pressure is measured before and after the revascularization procedure.

SECONDARY OUTCOMES:
WIfI stage | Pre-procedural, post-procedural (within 5 days) and 3 months after the index procedure
  Change in WIfI (wound, ischemia, foot infection) stage is documented before and after the revascularization procedure.
Rutherford category | Pre-procedural, post-procedural (within 5 days) and 3 months after the index procedure
  Change in Rutherford category is documented before and after the revascularization procedure.
Primary patency | Post-procedural (within 5 days) and 3 months after the index procedure
  Primary patency of the treated arterial lesion is documented after the procedure
Secondary patency | Post-procedural (within 5 days) and 3 months after the index procedure
  Secondary patency of the treated arterial lesion is documented after the procedure
Limb salvage | Post-procedural (within 5 days) and 3 months after the index procedure
  Limb salvage of the treated extremity is documented after the procedure
Ankle-brachial index (ABI) | Pre-procedural, post-procedural (within 5 days) and 3 months after the index procedure
  Change in ABI is documented before and after the revascularization procedure.
Fluorescence angiography | Pre-procedural, post-procedural (within 5 days) and 3 months after the index procedure
  Change in fluorescence angiography is documented before and after the revascularization procedure.
Survival | Post-procedural (within 5 days) and 3 months after the index procedure
  Survival of patients after the revascularization.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Vascular Surgery, Medical University Innsbruck, Innsbruck, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Halliday A, Bax JJ. The 2017 ESC Guidelines on the Diagnosis and Treatment of Peripheral Arterial Diseases, in Collaboration With the European Society for Vascular Surgery (ESVS). Eur J Vasc Endovasc Surg. 2018 Mar;55(3):301-302. doi: 10.1016/j.ejvs.2018.03.004. No abstract available. PMID 29579461
- [Background] Conte MS, Bradbury AW, Kolh P, White JV, Dick F, Fitridge R, Mills JL, Ricco JB, Suresh KR, Murad MH, Aboyans V, Aksoy M, Alexandrescu VA, Armstrong D, Azuma N, Belch J, Bergoeing M, Bjorck M, Chakfe N, Cheng S, Dawson J, Debus ES, Dueck A, Duval S, Eckstein HH, Ferraresi R, Gambhir R, Gargiulo M, Geraghty P, Goode S, Gray B, Guo W, Gupta PC, Hinchliffe R, Jetty P, Komori K, Lavery L, Liang W, Lookstein R, Menard M, Misra S, Miyata T, Moneta G, Munoa Prado JA, Munoz A, Paolini JE, Patel M, Pomposelli F, Powell R, Robless P, Rogers L, Schanzer A, Schneider P, Taylor S, De Ceniga MV, Veller M, Vermassen F, Wang J, Wang S; GVG Writing Group for the Joint Guidelines of the Society for Vascular Surgery (SVS), European Society for Vascular Surgery (ESVS), and World Federation of Vascular Societies (WFVS). Global Vascular Guidelines on the Management of Chronic Limb-Threatening Ischemia. Eur J Vasc Endovasc Surg. 2019 Jul;58(1S):S1-S109.e33. doi: 10.1016/j.ejvs.2019.05.006. Epub 2019 Jun 8. PMID 31182334
- [Background] Rutherford RB, Baker JD, Ernst C, Johnston KW, Porter JM, Ahn S, Jones DN. Recommended standards for reports dealing with lower extremity ischemia: revised version. J Vasc Surg. 1997 Sep;26(3):517-38. doi: 10.1016/s0741-5214(97)70045-4. PMID 9308598